CLINICAL TRIAL: NCT02968238
Title: Cognitive-behavioral Therapy Versus Yoga for the Treatment of Worry in Anxious Older Adults: A Randomized Preference Trial
Brief Title: Tranquil Moments II-CBT vs. Yoga for Worry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00041530; CER-1511-33007 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2019-12

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy; Yoga

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CBT preference arm (Active Comparator): CBT preference arm consists of participants who are randomized to the preference condition and choose to receive cognitive-behavioral therapy (CBT). CBT consists of 10 weeks of weekly treatment.
  Interventions: Behavioral: Cognitive-behavioral therapy
- Yoga preference arm (Active Comparator): Yoga preference arm consists of participants who are randomized to the preference condition and choose to receive yoga. Yoga consists of 10 weeks of bi-weekly treatment (total = 20 treatments).
  Interventions: Behavioral: Yoga
- CBT randomized arm (Active Comparator): CBT randomized arm consists of participants who are randomized to the random condition and are randomized to receive cognitive-behavioral therapy (CBT). CBT consists of 10 weeks of weekly treatment.
  Interventions: Behavioral: Cognitive-behavioral therapy
- Yoga randomized arm (Active Comparator): Yoga randomized arm consists of participants who are randomized to the random condition and are randomized to receive yoga. Yoga consists of 10 weeks of bi-weekly treatment (total = 20 treatments).
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — 10 weekly sessions of cognitive-behavioral therapy
  Other Names: CBT
  Arms: CBT preference arm; CBT randomized arm
Behavioral: Yoga — 10 weeks of biweekly yoga sessions (N = 20)
  Arms: Yoga preference arm; Yoga randomized arm

SUMMARY:
Anxiety disorders are the most prevalent psychiatric disorders. Among older adults, anxiety is more common that depression, yet research on the nature and treatment of anxiety has lagged far behind that of depression. The investigators' work has demonstrated that CBT is superior to enhanced usual care as well as supportive therapy in improving worry, depressive symptoms, and sleep, and these improvements are maintained for up to 1 year upon completing treatment. Research demonstrates that yoga reduces anxiety symptoms and the investigators' own work demonstrates that yoga improves sleep. However, no one has conducted a comparative effectiveness trial of CBT and yoga for treating worry in older adults. In fact, there are very few comparative effectiveness trials for treating late-life anxiety. Thus, clinicians are unable to provide an informed recommendation of one treatment over the other. The investigators propose a two-stage randomized preference trial comparing 1) cognitive-behavioral therapy with 2) yoga for the treatment of worry in a sample of older adults. Participants will be randomized to either the preference group (participants choose the treatment) or to the random group (participants are randomized to 1 of the 2 treatments). This study design allows for the calculation of traditional treatment effects (differences in outcomes between participants randomized to either CBT or yoga), selection effects (differences in outcomes between participants who choose CBT and those who choose yoga), and preference effects (differences in outcomes between participants who choose their treatment and those who are randomized to treatment).

DETAILED DESCRIPTION:
The primary aim of this study is to compare the effects of CBT and yoga on worry in older adults (as assessed by the PSWQ-A measured at post-intervention, Week 11). Secondary aims are to compare the effects of these treatments on anxiety and sleep (as assessed by the PROMIS anxiety scale and the ISI, respectively, measured at post-intervention, Week 11). Exploratory aims are to determine participant preference for CBT vs. yoga; examine participant preference effects on worry, anxiety, sleep, adherence to treatment, and attrition rates; and examine selection effects on worry, anxiety, sleep, adherence to treatment, and attrition rates. All analyses will be repeated for measures assessed at Week 37.

The treatment effect for the primary aim will be estimated by comparing mean PSWQ-A scores between CBT and yoga groups in the random group (N=250, 125 per group) using constrained mixed-model repeated measures analysis of covariance with an unstructured covariance matrix to account for the fact that the multiple measurements (at baseline-Week 0, mid-intervention-Week 6, post-intervention-Week 11) from participants are not independent. The model will contain terms for baseline psychotropic medication use, gender and race (both related to depression), and intervention effects that are specific to each follow-up time. Because this arm of the trial has been randomized, we will constrain the pre-randomization intervention-specific outcome means to be the same. A contrast will be used to test the primary hypothesis at the post-intervention (Week 11) time point using a two-sided 0.05 significance level. In the primary analysis, all randomized participants will be included in their original study group for analysis regardless of the final mode of intervention or the extent of compliance with the study protocol; that is, the primary analysis will follow an "intent to treat" philosophy.

As part of the secondary aims, the estimation of selection and preference effects will be performed with mixed models based on the complete sample using data collected in both preference and randomized arms of the trial. Therefore, these analyses will be based on a sample size of 500 individuals. The adjusted means and variance-covariance matrix needed to compute these effects and their standard error will be estimated from the fitted model. The standard error associated with the preference and selection effects will be derived using the delta-method and/or a bootstrapping approach, as needed.

Consistency of intervention effects will be explored within the following baseline subgroups: 1) depressive symptoms from PROMIS measure (none or mild vs. moderate or severe), 2) use of psychotropic meds (any vs none), 3) age (60-79 vs 80+), 4) gender (female/male), and 5) race (White vs. other races).

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and older
* Moderate to severe levels of worry

Exclusion Criteria:

* Currently receiving psychotherapy
* Currently practicing yoga
* Active alcohol/substance abuse
* Dementia
* Current psychotic symptoms
* Active suicidal ideation with plan and intent
* Hearing loss that would prevent a person from participating in telephone/class sessions

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Penn State Worry Questionnaire-Abbreviated | Week 11
  worry symptoms

SECONDARY OUTCOMES:
PROMIS Anxiety | Week 11, Week 37
  anxiety symptoms
Insomnia Sleep Index | Week 11, Week 37
  sleep problems
Penn State Worry Questionnaire-Abbreviated | Week 6, Week 37
  worry symptoms
PROMIS 29 | Week 11, Week 37
  29-item self-report measure with 4 items each for the following: physical function, anxiety, depression, fatigue, sleep, social function, pain interference; 1 item for average pain intensity
PROMIS Depression | Week 11, Week 37
  depressive symptoms
PROMIS Physical Function with Mobility Aid | Week 11, Week 37
  Self-report measure of current capability for physical activities
GAD-7 | Week 11, Week 37
  Self-report symptoms of Generalized Anxiety Disorder
Cornell Medical Services Index | Week 11, Week 37
  measure of medical care utilization
Client Satisfaction Questionnaire | Week 11
  self-report measure of satisfaction with treatment
Working Alliance Inventory, Client and Therapist | Week 11, Week 37
  assesses therapist-patient working alliance; measures are completed by the participant and the therapist
Adherence to the intervention as assessed by the number of sessions attended | Week 11
  adherence to treatment
Attrition from the intervention as assessed by the number of participants who do not complete study assessments at Week 11 and Week 37 | Week 11, Week 37
  attrition from study
FES-I | Week 11, Week 37
  falls self-efficacy
Falls | Week 11, Week 37
  self-report incidence of falls
Penn State Worry Questionnaire-Abbreviated | Week 37
  worry symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Brenes, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danhauer SC, Miller ME, Divers J, Anderson A, Hargis G, Brenes GA. Long-Term Effects of Cognitive-Behavioral Therapy and Yoga for Worried Older Adults. Am J Geriatr Psychiatry. 2022 Sep;30(9):979-990. doi: 10.1016/j.jagp.2022.02.002. Epub 2022 Feb 6. PMID 35260292
- [Derived] Sohl SJ, Brenes GA, Krucoff C, Hargis G, Anderson A, Miller ME, Danhauer SC. Ensuring Yoga Intervention Fidelity in a Randomized Preference Trial for the Treatment of Worry in Older Adults. J Altern Complement Med. 2021 Jun;27(6):489-495. doi: 10.1089/acm.2020.0476. Epub 2021 Mar 8. PMID 33684325
- [Derived] Brenes GA, Divers J, Miller ME, Danhauer SC. A randomized preference trial of cognitive-behavioral therapy and yoga for the treatment of worry in anxious older adults. Contemp Clin Trials Commun. 2018 May 4;10:169-176. doi: 10.1016/j.conctc.2018.05.002. eCollection 2018 Jun. PMID 30009275

DOCUMENTS (1):
  • Informed Consent Form (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT02968238/ICF_000.pdf